CLINICAL TRIAL: NCT00000795
Title: A Phase I Safety and Immunogenicity Trial of UBI Multivalent HIV-1 Peptide Immunogen in HIV-1 Seronegative Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 017
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2002-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: HIV-1 Peptide Immunogen, Multivalent

SUMMARY:
To evaluate, in healthy adult volunteers, the safety and immunogenicity of multivalent HIV-1 peptide immunogen, a formulation of HIV-1 gp120 principal neutralizing domain (PND) branched synthetic peptides from 15 viral strains representative of diverse worldwide isolates.

Because there is considerable variation among HIV-1 virus strains from differing geographical locations worldwide, a multivalent peptide vaccine has been constructed to include prevalent and divergent isolates, potentially providing for wide coverage of geographically isolated epidemics.

DETAILED DESCRIPTION:
Because there is considerable variation among HIV-1 virus strains from differing geographical locations worldwide, a multivalent peptide vaccine has been constructed to include prevalent and divergent isolates, potentially providing for wide coverage of geographically isolated epidemics.

Fourteen volunteers are entered at one of two dose levels of multivalent candidate vaccine. At each dose level, 12 volunteers receive vaccine and two receive placebo. At least eight volunteers at the low dose level must be monitored for 2 weeks before subsequent volunteers are entered at the high dose. Intramuscular injections are given on days 0, 28, and 168, and patients are followed for a minimum of 48 weeks after the initial immunization. Approximately 13 clinical visits are required.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* HIV negativity by ELISA within 8 weeks of immunization.
* CD4 count >= 400 cells/mm3.
* Normal urinalysis.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Positive hepatitis B surface antigen.
* Medical or psychiatric condition or occupational responsibilities that preclude study compliance.
* Active syphilis. NOTE: Subjects whose serology is documented to be a false positive or due to a remote (> 6 months) treated infection are eligible.
* Active tuberculosis. NOTE: Subjects with a positive PPD and normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy are eligible.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, or autoimmune disease.
* History of anaphylaxis or other serious reactions to vaccines.

Prior Medication:

Excluded:

* History of immunosuppressive medications.
* Live attenuated vaccines within 60 days prior to study entry (NOTE: Medically indicated subunit or killed vaccines, e.g., influenza or pneumococcal, are not exclusionary, but should not be given within 2 weeks of HIV immunization).
* Experimental agents within 30 days prior to study entry.
* Prior HIV vaccines.

Prior Treatment:

Excluded:

* Blood products or immunoglobulin within the past 6 months.

Identifiable higher risk behavior for HIV infection, including the following:

* History of injection drug use within the past 12 months.
* Higher risk sexual behavior as defined by the AVEG.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28

CONTACTS AND LOCATIONS:
Overall Officials: Keefer M, Study Chair
Locations (1):
- Johns Hopkins Univ / Ctr for Immunological Research, Baltimore, Maryland, United States

REFERENCES:
- [Background] Kelleher AD, Emery S, Cunningham P, Duncombe C, Carr A, Golding H, Forde S, Hudson J, Roggensack M, Forrest BD, Cooper DA. Safety and immunogenicity of UBI HIV-1MN octameric V3 peptide vaccine administered by subcutaneous injection. AIDS Res Hum Retroviruses. 1997 Jan 1;13(1):29-32. doi: 10.1089/aid.1997.13.29. PMID 8989424
- [Background] Evans TG, Fitzgerald T, Gibbons DC, Keefer MC, Soucier H. Th1/Th2 cytokine responses following HIV-1 immunization in seronegative volunteers. The AIDS Vaccine Evaluation Group. Clin Exp Immunol. 1998 Feb;111(2):243-50. doi: 10.1046/j.1365-2249.1998.00486.x. PMID 9486388
- [Background] Kahn J, Murcar N, Elbeik T, Staprans S, Hanson C, Mayer Y, Doyle R, Gonzalez L, Koff W. UBI HIV-1MN octameric V3 peptide vaccine in HIV-1 negative humans. Conf Adv AIDS Vaccine Dev. 1996 Feb 11-15:167 [Poster 47]